CLINICAL TRIAL: NCT00399113
Title: An Open-Label Phase I Safety, Pharmacokinetic & Dosimetry Study of 188Re-PTI-6D2 in Patients With Metastatic Melanoma
Brief Title: Safety Study of 188Re-PTI-6D2 in Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pain Therapeutics (Industry)
Responsible Party: Michael R. Marsman, PharmD, Pain Therapeutics, Inc.
Organization: PainT (Unknown)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTI-6D2-A
Record Dates: First submitted 2006-11-13; First posted 2006-11-14 (Estimated); Last update posted 2011-07-14 (Estimated); Status verified 2011-07

CONDITIONS: Metastatic Melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: 188Re-PTI-6D2 — monoclonal antibody

SUMMARY:
The purpose of this first-in-man study is to evaluate the safety of 188Re-PTI-6D2 in patients with metastatic melanoma. All patients will receive a tracer dose of 188Re-PTI-6D2 in order to provide information on how the monoclonal antibody is distributed throughout the body and to assess tumor targeting. No therapeutic dose of radiation will be given in the first study.

DETAILED DESCRIPTION:
This study will evaluate the safety and feasibility of the administration of 188Re-PTI-6D2 in patients with metastatic melanoma. Patients with confirmed Stage IIIc (unresectable) or Stage IV melanoma who meet all eligibility criteria will undergo a thorough physical examination and baseline tumor imaging (whole body 18FDG PET/CT and MRI brain) to document all sites of tumor.

Treatment will be administered on an inpatient basis. An initial cohort of 3 patients will receive a tracer dose of 188Re-PTI-6D2 without any preceding unlabeled antibody. The tracer dose will consist of 10 mCi of rhenium-labeled antibody; the amount of antibody (in mg) will depend on specific activity and is estimated to range from 2 to 10 mg. Additional cohorts of three patients each will receive 10 mg, 20 mg, and 50 mg of unlabeled PTI-6D2 immediately preceding administration of the tracer dose. Patients will undergo serial gamma scans and SPECT/CT imaging at specified time points. Blood samples will be obtained prior to dosing and at specified intervals for PK measurements of the mAb as well as for measurement of serum radioactivity. Urine will also be collected for all patients to measure excreted radioactivity. Patients will be closely monitored for safety throughout the duration of the study.

Patients will remain at the study center for 48 hours after infusion to allow adequate time for post-treatment safety observation, monoclonal antibody clearance and rhenium decay. Prior to the escalation of the dose of unlabeled PTI-6D2, safety data from the inpatient period and 2-week follow-up visit for the three patients at the current dose level will be reviewed. If there is no evidence of a safety risk, the dose of unlabeled PTI-6D2 will be escalated for the next cohort of patients. Dose escalation of unlabeled antibody will occur according to a specific scheme.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed Stage IIIc (unresectable) or Stage IV metastatic melanoma;
* measurable disease;
* at least 18 years of age;
* Karnofsky status at least 50%;
* life expectancy > 3 months;
* at least 4 weeks since prior therapy;
* adequate organ and marrow function defined by screening laboratory tests;
* negative screening human anti-murine antibodies;
* females of child-bearing potential must be practicing an acceptable method of birth control and have a negative urine pregnancy test;
* written informed consent obtained

Exclusion Criteria:

* Chemotherapy or radiation therapy within 4 weeks or poor recovery from therapy > 4 weeks ago;
* investigational drug within 30 days;
* brain metastasis (all patients must have contrast-enhanced MRI within 2 weeks of treatment to rule out);
* ocular inflammatory disease or ocular neoplasm (all patients must have fundoscopic and slit lamp examination within 2 weeks of treatment to rule out exclusionary ocular pathology);
* prior parenteral exposure to murine proteins;
* positive hep B surface Ag, hep C antibody, or HIV test at screening;
* uncontrolled intercurrent illness;
* pregnant/breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2007-05; Primary Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
To select the amount of unlabeled PTI-6D2 to administer immediately prior to a tracer dose of 188Re-PTI-6D2 in order to achieve preferred tumor targeting
To generate pharmacokinetic (PK) and biodistribution data of 188Re-PTI-6D2 in patients with metastatic melanoma in order to estimate radiation doses absorbed to tumor and critical organs
To determine the frequency of HAMA response associated with 188Re-PTI-6D2 administration

CONTACTS AND LOCATIONS:
Overall Officials: Eithan Galun, M.D., Principal Investigator — Hadassah Hebrew University Hospital; Jacob Schachter, M.D., Principal Investigator — Chaim Sheba Medical Center; Tzila Zwas, M.D., Principal Investigator — Chaim Sheba Medical Center
Locations (2):
- Israel (2):
  - Hadassah Hebrew University Hospital, Jerusalem
  - Chaim Sheba Medical Center, Tel Litwinsky